CLINICAL TRIAL: NCT05693324
Title: Minority Joy and Minority Stress in Trans People: an Intervention Study Including a Longitudinal Mapping of Health Factors
Brief Title: Minority Joy and Minority Stress in Trans People: an Intervention Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Ida Flink, Assistant professor, Örebro University, Sweden
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: JoyStressIntervention
Record Dates: First submitted 2023-01-10; First posted 2023-01-23 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Emotional Problem; Pain, Back; Quality of Life
Keywords: transpeople; minority joy; minority stress
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Intervention Model Description: This study employs a single-case experimental design with randomized waiting period lengths (4, or 6 weeks) as well as randomization to three treatment arms (same content, different progress through the three modules). Included in the design is also standardized pre- and post measurement allowing for single group analysis of change. In addition, we collect qualitative data from participants, detailing how the intervention is experienced.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 1 Minority stress (Active Comparator): Intervention starts with the minority stress module, followed by worry and then compassion.
  Modules are given with a trans-affirmative stance, based on the minority stress model. The minority stress module contains psychoeducation on minority stress and minority joy as well as behavioral interventions. The worry module contains cognitive interventions. The compassion module targets internalized transphobia and is based on compassion-focused therapy.
  Interventions: Behavioral: Minority stress
- 2 Minority stress (Active Comparator): Intervention starts with minority stress module, followed by compassion and then worry.
  Modules are given with a trans-affirmative stance, based on the minority stress model. The minority stress module contains psychoeducation on minority stress and minority joy as well as behavioral interventions. The worry module contains cognitive interventions. The compassion module targets internalized transphobia and is based on compassion-focused therapy.
  Interventions: Behavioral: Minority stress
- 3 Worry (Active Comparator): Intervention starts with worry module, followed by minority stress and then compassion.
  Modules are given with a trans-affirmative stance, based on the minority stress model. The minority stress module contains psychoeducation on minority stress and minority joy as well as behavioral interventions. The worry module contains cognitive interventions. The compassion module targets internalized transphobia and is based on compassion-focused therapy.
  Interventions: Behavioral: Minority stress
- 4 Worry (Active Comparator): Intervention starts with worry module, followed by compassion and then minority stress.
  Modules are given with a trans-affirmative stance, based on the minority stress model. The minority stress module contains psychoeducation on minority stress and minority joy as well as behavioral interventions. The worry module contains cognitive interventions. The compassion module targets internalized transphobia and is based on compassion-focused therapy.
  Interventions: Behavioral: Minority stress
- 5 Compassion (Active Comparator): Intervention starts with compassion module, followed by minority stress and then worry.
  Modules are given with a trans-affirmative stance, based on the minority stress model. The minority stress module contains psychoeducation on minority stress and minority joy as well as behavioral interventions. The worry module contains cognitive interventions. The compassion module targets internalized transphobia and is based on compassion-focused therapy.
  Interventions: Behavioral: Minority stress
- 6 Compassion (Active Comparator): Intervention starts with compassion, followed by worry and then minority stress.
  Modules are given with a trans-affirmative stance, based on the minority stress model. The minority stress module contains psychoeducation on minority stress and minority joy as well as behavioral interventions. The worry module contains cognitive interventions. The compassion module targets internalized transphobia and is based on compassion-focused therapy.
  Interventions: Behavioral: Minority stress

INTERVENTIONS:
Behavioral: Minority stress — Intervention based on Cognitive Behavioural and Compassion Focused Treatments
  Other Names: Worry; Compassion

SUMMARY:
The aim of this project is to get a better understanding of transgender and gender non-conforming (TGNC) people's experiences of minority joy and minority stress over time. Further, the project explores how these experiences covary with psychiatric and physical ill health and quality of life before, during and after a TGNC affirmative intervention in adult and adolescent participants over 15 years of age. The intervention consists of three parts, given in randomized order: 1. Psychoeducation and behavioral interventions about external minority stress, 2. Cognitive interventions targeting worry, and 3. Self-compassion aiming to relieve internalized transphobia.

This project uses a mixed methods data collection consisting of interviews as well as a replicated single case design (SCED). More detailed pre- and post measurements will also be collected. The interviews enable us to explore minority joy in detail, as well as getting feedback about the feasibility and acceptability of the intervention. The SCED enables us to visualize the interplay between everyday experiences and health, while testing the affirmative program. The project will provide much needed knowledge, which in turn will improve health in TGNC people.

DETAILED DESCRIPTION:
The aim of this project is to exploratively investigate TGNC people's experiences of minority joy, and to get a better understanding of their experiences of minority joy and minority stress over time. Further, the project aims to explore how these experiences covary with psychiatric and physical ill health and quality of life before, during and after a TGNC affirmative intervention in adult and adolescent participants over 15 years of age. The intervention targets minority stress and consists of three parts, given in randomized order: 1. Psychoeducation about external minority stress including behavioral interventions, 2. Cognitive interventions targeting worry, and 3. Self-compassion interventions aiming to relieve internalized transphobia.

This project is designed to collect data on external minority stress and minority joy over time and at the same time to test an intervention based on the minority stress model, targeting internal minority stress, worry, and self-compassion. This is done using a replicated single case design, which makes it possible to visualize the interplay between everyday experiences and health in a number of individuals. It also tests an affirmative program targeting factors that have been suggested as important in the development of ill health in minority populations. This is done in a way that allows visualizing change directly, giving an opportunity for direct feedback and adaptation, providing an understanding of the interplay between minority stress, minority joy and health. It will also allow us to visualize the potential of the separate parts of the intervention, as well as the intervention as a whole, including feasibility and how it is experienced by participants.

To allow us to tap into a variability of experiences, both TGNC people doing well and TGNC people reporting some health problems will be recruited (about 35 each). The preventative effect of the intervention will therefore also be investigated, mainly qualitatively as part of the evaluation of the intervention.

Research questions:

1. How often and in which situations do TGNC people with and without symptoms of health problems experience minority stress and minority joy over time?
2. How do minority stress and minority joy covary with physical and psychological health (pain, anxiety, and depression) and quality of life over time in TGNC people with and without symptoms of health problems?
3. How do minority stress and minority joy covary with suggested mediators (worry, self-compassion) over time in TGNC people with and without symptoms of health problems?
4. Does a TGNC affirmative intervention targeting minority stress, worry, and self-compassion influence health and quality of life in TGNC people with health problems, and are there distinct differences regarding the three modules?
5. How feasible is the intervention, and how is it experienced by participants with and without health problems?

The project consists of a mixed methods data-collection. Data-collection for aims one, two, three and four will consist of a single case experimental design with repeated weekly measurements, including longer pre- and post measurements. Research question five will use answers from the post-measurements as well as semi-structured interviews held with participants after the intervention.

Data collection

1. SCED with repeated measurements, including pre- and post measurements In a SCED, several participants fill in repeated measurements, during periods of intervention (Phase B) and no intervention (Phase A). In this case, participants fill in measurements weekly for a maximum of 24 weeks starting with a 4- or 6-weeks randomized baseline followed by three separate intervention modules. After and between the intervention modules there are three weeks of data collection without any active intervention. Thus, the data-collection includes periods where life is observed interspersed with weeks where individuals learn new skills and are supported by a therapist with an affirmative stance.

Before baseline and after the intervention, longer questionnaires will be filled in to get detailed information about our participants, and to enable us to relate validated questionnaires to the questions used for the weekly repeated measurements. It also allows the use of some more standard statistical analyses. The single case experimental design study (SCED) has several aims and is collecting weekly data over a period of 22-24 weeks.

The weekly questionnaire that will be developed specifically for the data collection includes two to three items about each area (depression, anxiety, musculoskeletal pain, self-compassion, worry, quality of life, minority joy, minority stress). This will result in 20 questions that focus on:

1. How and where minority stress and minority joy are experienced on a weekly basis
2. How intervention targets (self-compassion and worry) as well as symptoms (anxiety, depression, and musculoskeletal pain) and quality of life vary over time.

There will also be a weekly open question where participants can describe a specific experience of minority stress or joy or comment on the intervention.

The baseline, breaks and follow-up period enable us to separate the intervention modules more clearly from each other, which makes it possible to relate changes to the start or end of an intervention module, strengthening the external validity of the study. The different sequences of modules result in six different arms that participants will be randomized to (in blocks of six) and enable us to see if outcome seems to be more dependent on time or on content. Here, the first B-phase will be the most informative, since the intervention given first is the least influenced by content in the other modules.

Pre- and post-measurements (collected at the start of baseline and just after the last intervention module) enable us to collect full measurements on self-compassion, worry, and outcome variables, which enables us to relate validated measurements to the scores on the items on our weekly measurements and do simple pre-post comparisons (more advanced analyses will likely not be possible due to power issues). Also, detailed demographic information will be collected before the intervention to be able to describe participants' living conditions. After the intervention, questions about feasibility and agreeableness of the intervention are added.

2. Semi structured interviews about feasibility and participant's experience of intervention After the intervention participants with and without symptoms of health problems will be asked if they are interested to take part in an interview about the intervention. Here, detailed information can be collected about how the intervention was experienced, what was missing, which modules were felt to be the most helpful and if there were any negative effects. It will also be possible to let participants express if, how, and where they would like to receive similar interventions in the future. Of specific interest is how participants without or with low levels of symptoms of health problems experienced the intervention, which could give us an idea about its preventative potential.

ELIGIBILITY:
Inclusion Criteria:

* Identity other than assigned sex at birth
* Access to internet and ability to fill in questionnaires in Swedish

Exclusion Criteria:

* Ongoing psychiatric or other problems that make it unlikely that intervention schedule can be followed (e.g. acute problems requiring other care, inability to schedule sessions)

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — A gender identity different from assigned sex at birth
Enrollment: 70 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Weekly measurement, specifically constructed for this study | 20-24 weeks
  Assesses minority stress/joy, self-compassion, worry, pain, depression, anxiety, and quality of life with two questions each, resulting in 16 short questions, answerable between 1-10. For self-compassion, minority joy and quality of life, higher scores indicate better functioning, for depression, minority stress, anxiety, pain, worry, higher scores indicate more problems. Additionally, experiences can be described in a free text.

SECONDARY OUTCOMES:
Self compassion scale | pre- and post measurement with 20-24 weeks between measurements, collected at the start of baseline and just after the last intervention module
  12 questions indicating ability to feel self-compassion and act in a self-compassionate way. Scores range from 1-5 with total scores of 60. Higher scores indicate better functioning in regards to having self-compassion.
Penn State Worry questionnaire | pre- and post measurement with 20-24 weeks between measurements, collected at the start of baseline and just after the last intervention module
  Worry is assessed with 9 items scoring between 1-5 with total scores of 45. Higher scores indicate more worry.
Pain grades | pre- and post measurement with 20-24 weeks between measurements, collected at the start of baseline and just after the last intervention module
  Pain duration, intensity and function are combined in 5 pain grades (0, I, II, III, IV), where pain problems (grades III and IV) are indicated if pain is experienced at least every month and function is impaired at least somewhat in one of the three areas work, social contacts or leisure time.
Depression Anxiety Stress Scale, DASS | pre- and post measurement with 20-24 weeks between measurements, collected at the start of baseline and just after the last intervention module
  Measures symtoms of depressin, anxiety and stress in three subscales of 7 items each (total 21 items). Each item scores between 0-3, with each subscale scoring between 0-21, with higher scores indicating more problems.
quality of life, SWLS | pre- and post measurement with 20-24 weeks between measurements, collected at the start of baseline and just after the last intervention module
  Quality of life is assessed with the SWLS, including five items, answerable on a scale from 1-7 with total scores between 5-35. Higher scores indicate higher quality of life.
Gender Identity Microaggression Scale, GIMS | pre- and post measurement with 20-24 weeks between measurements, collected at the start of baseline and just after the last intervention module
  14 items with concrete situations, such as misgendering, that participant can indicate if they have experienced or not.

CONTACTS AND LOCATIONS:
Overall Officials: Matilda Wurm, PhD, Principal Investigator — Örebro University, Sweden
Locations (1):
- Örebro University, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No
Data will not be shared freely, but will be saved on the university server. Access can be requested by contacting PI or data manager at the university.